CLINICAL TRIAL: NCT02213367
Title: Phase 3 Study, Exploratory, Disease Activity Controlled Dose Escalating Study to Assess the Efficacy, and Safety of Treatment With Bilastine 20 mg, 40 mg and 80 mg in Chronic Spontaneous Urticaria.
Brief Title: Bilastine Updosing in Chronic Spontaneous Urticaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, K. Weller, PD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUCSU
Record Dates: First submitted 2014-08-08; First posted 2014-08-11 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — bilastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 20 mg Bilastin (Active Comparator): 20mg Bilastine once daily
  Interventions: Drug: Bilastine; Drug: Bilastin
- Bilastin 40mg (Active Comparator): 40 mg Bilastine once daily, intake of two tablets 20mg Bilastine
  Interventions: Drug: Bilastine; Drug: Bilastin
- Bilastin 80mg (Active Comparator): 80 mg Bilastine once daily, intake of four tablets 20mg Bilastine
  Interventions: Drug: Bilastine; Drug: Bilastin

INTERVENTIONS:
Drug: Bilastine — 20mg (8 weeks)
  Other Names: Bilaxten
Drug: Bilastine — 40mg
  Other Names: Bilaxten
Drug: Bilastin — 80mg
  Other Names: Bilaxten

SUMMARY:
Chronic spontaneous urticaria (CSU), formerly also known as chronic idiopathic urticaria and chronic urticaria (CU), is one of the most frequent skin diseases. At any time, 0.5-1% of the population suffers from the disease. Although all age groups can be affected, the peak incidence is seen between 20 and 40 years of age. The duration of the disease is generally several years but is likely to be longer in more severe cases, cases with concurrent angioedema, in combination with physical urticaria or with a positive autologous serum skin test (autoreactivity). CSU has major detrimental effects on quality of life, with sleep deprivation and psychiatric comorbidity being frequent. It also has a large impact on society in terms of direct and indirect health care costs as well as reduced performance at work and in private life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years and older
* History of active chronic spontaneous urticaria with or without associated angioedema for at least three days per week over the last 6 weeks prior to visit 1. - Urticaria symptoms must comprise wheals and itch
* History of failed treatment with an antihistamine other than bilastine in standard (licensed) dose.
* UAS7 of ≥14 during baseline
* Informed consent signed and dated
* Able to read, understand and willing to sign the informed consent form and abide with study procedures
* Willing, committed and able to return for all clinic visits and complete all study-related procedures
* In females of childbearing potential: negative pregnancy test; females willing to use highly effective contraception (Pearl-Index < 1) a woman will be considered not of childbearing potential if she is post-menopausal for > 2 years or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy)
* No participation in other clinical trials 4 weeks before and after participation in this study

Exclusion Criteria:

* Chronic spontaneous urticaria patients with a known resistance to bilastine
* Isolated presence or domination of inducible forms of urticaria or cholinergic urticaria (no chronic spontaneous urticaria)
* History of adverse reactions to bilastine or known hypersensitivity to bilastine or its ingredients
* Intake of oral corticosteroids or intravenously applied corticosteroids within 28 days prior to screening visit
* Use of depot corticosteroids within 3 months prior to screening visit (inhaled corticosteroids are allowed)
* Use of systemic immunosupressants/immunomodulators such as ciclosporin, dapsone, metotrexate, and comparable drugs within 28 days prior to screening visit.
* Use of UV-therapy within 28 days prior to visit 1
* Significant medical condition, in the opinion of the Investigator, rendering the patient immunocompromised or not suitable for a clinical trial
* Significant concomitant illness, in the opinion of the Investigator, that would adversely affect the subject's participation or evaluation in this study
* ECG alterations of repolarisation (QTc prolongations >450ms or increase of QTc >60ms as compared to the baseline assessment)
* Blood pressure >180/100 mmHg and/or heart rate >100/min
* Evidence of significant hepatic or renal disease (GOT and/or GPT >2 times above the upper reference value, serum creatinine 1.5 times above the upper reference value)
* Subjects for whom there is concern, in the opinion of the Investigator, about compliance with the protocol procedures
* The presence of a permanent gastrointestinal condition which may influence the oral therapy (chronic diarrhoea diseases, congenital malformations or surgical mutilations of gastrointestinal tract)
* Presence of active cancer which requires chemotherapy or radiation therapy
* Presence of alcohol abuse or drug addiction
* Pregnancy or breast-feeding
* Subjects who are inmates of psychiatric wards, prisons, or other state institutions. Existing or planned placement in an institution after ruling according to § 40 passage 1, number 4 AMG (Arzneimittelgesetz).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Effects of standard dose (20 mg) and higher than standard dose of bilastine (40 mg and 80 mg) on disease activity in patients with chronic spontaneous urticaria. | 8 weeks

SECONDARY OUTCOMES:
To assess the effects of standard dose (20 mg) and higher than standard dose of bilastine (40 mg and 80 mg) on quality of life impairment in patients with chronic spontaneous urticaria. | 4 weeks
  To assess the safety of bilastine in doses of 20 mg, 40 mg and 80 mg in chronic spontaneous urticaria patients by documentation of adverse events.
  To assess the effects of standard dose (20 mg) and higher than standard dose of bilastine (40 mg and 80 mg) on biomarkers of chronic spontaneous urticaria, such as substance P and D-Dimers

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Weller, MD, Principal Investigator — Dpt. of Dermatology and Allergy , Charité
Locations (1):
- Dpt. of Dermatology and Allergy, Berlin, Germany, Germany